CLINICAL TRIAL: NCT03274336
Title: Influence of Audiovisual Aids in the Preanesthetic Interview: A Comparison of the Effect of Face-to-face-interview Versus a Brochure and Video Assisted Interview
Brief Title: Influence of Audiovisual Aids in the Preanesthetic Interview
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Schulthess_Anä_12
Record Dates: First submitted 2017-08-19; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Patient Satisfaction
Keywords: patient satisfaction; preanesthesia; movie; brochure; face-to-face interview
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires; Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interview (Active Comparator): questionnaire after face-to-face interview
  Interventions: Behavioral: questionnaire; Behavioral: face-to-face interview; Behavioral: brochure; Behavioral: movie
- brochure (Placebo Comparator): questionnaire interview plus brochure
  Interventions: Behavioral: questionnaire; Behavioral: brochure
- movie (Placebo Comparator): questionnaire interview plus movie
  Interventions: Behavioral: questionnaire; Behavioral: movie

INTERVENTIONS:
Behavioral: questionnaire — questionnaire post preanesthetic interview
Behavioral: face-to-face interview — Group A = face-to-face interview
  Arms: interview
Behavioral: brochure — after reading a brochure a face to face interview will take place
  Arms: brochure; interview
Behavioral: movie — after seeing a film about the procedure a face-to-face interview will take place
  Arms: interview; movie

SUMMARY:
1000 patients will be asked to fill out a questionnaire about preanesthetic visit right after the interview. On a daily randomization the Groups will be assigned to: Group A = face-to-face interview; Group B = interview plus brochure, Group C= interview plus movie.

Evaluation of patient satisfaction und knowledge transfer will be evaluated with a questionnaire filled out right after the interview with the anesthesist.

ELIGIBILITY:
Inclusion Criteria:

* voluntary

Exclusion Criteria:

* language Problems
* not able to read or write
* patients does not want to fill out questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1172 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction on a questionnaire | 15 Minutes
  Patient satisfaction after the preanesthetic interview is measured

SECONDARY OUTCOMES:
time | 30 Minutes
  time needed for the preanesthetic interview in Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Moser, MD, Principal Investigator — Schulthess Klinik